CLINICAL TRIAL: NCT05105750
Title: A Comparative Study on Antiplatelet Efficacy of Indobufen and Aspirin in Patients With Coronary Atherosclerosis
Brief Title: A Comparative Study of Indobufen and Aspirin in Patients With Coronary Atherosclerosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Dr., MD, Ph.D, Director of CCU Ward, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 016
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-10

CONDITIONS: Coronary Atherosclerosis
Keywords: Light Transmittance Aggregometry; Indobufen; Aspirin; Plasma Thromboxane; Urine 11-dehydro thromboxane
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; indobufen; BID protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin 100 mg/d therapy (Active Comparator)
  Interventions: Drug: aspirin 100 mg/d
- indobufen 200 mg bid therapy (Experimental)
  Interventions: Drug: indobufen 200 mg bid

INTERVENTIONS:
Drug: aspirin 100 mg/d — 100mg aspirin for at least 3 days followed by aspirin 100 mg/d
  Arms: aspirin 100 mg/d therapy
Drug: indobufen 200 mg bid — 100mg aspirin for at least 3 days followed by indobufen 200 mg bid
  Arms: indobufen 200 mg bid therapy

SUMMARY:
In addition, studies have found that indobufen can inhibit coagulation function in rats. Compared with aspirin, the duration of antiplatelet efficacy of indobufen was shorter, and the platelet function recovered completely 24 hours after drug withdrawal. However, there are few studies on the antiplatelet efficacy of indobufen. The investigators' previous study found that the inhibitory effect of indobufen 100 mg Bid on COX system in atherosclerosis or healthy volunteers was equivalent to that of aspirin 100 mg QD, but the inhibitory effect on platelet COX-1 channel was significantly weaker than that of aspirin 100 mg QD. In view of this, this study intends to investigate the antiplatelet effect of indobufen 200 mg Bid in patients with coronary atherosclerosis by comparing it with conventional-dose aspirin 100 mg QD.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of coronary atherosclerosis without indications for stent implantation.
2. Age ≥ 18 years, ≤ 65 years
3. Sign informed consent

Exclusion Criteria:

1. A history of asthma or allergic constitution or known allergy to indobufen or aspirin.
2. High risk of bleeding (low hemoglobin 10g / L, history of peptic ulcer disease, fecal occult blood positive or known active bleeding, history of cerebral hemorrhage within 6 months, history of fundus hemorrhage, etc).
3. Creatinine was 1.2 times higher than the upper limit of normal value and ALT was 1.2 times higher than the normal value.
4. History of smoking and alcoholism.
5. History of diabetes.
6. Pregnancy and lactation women.
7. Nonsteroidal anti-inflammatory or other antithrombotic drugs other than indobufen are required.
8. Any other reason may affect the results of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
MPA | Within 24 hours after one month of medication
  Maximum platelet aggregation induced by arachidonic acid
TXB2 | Within 1 month after one month of medication
  Plasma thromboxaneB2
11-dh-TXB2 | Within 1 month after one month of medication
  Urine 11-dehydro thromboxaneB2

SECONDARY OUTCOMES:
Adverse Events | Within 1 month after the first medication
  Monitor the bleeding events of subjects during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No